CLINICAL TRIAL: NCT00101413
Title: A Phase II Multicenter Uncontrolled Trial of BAY43-9006 in Patients With Relapsed or Refractory Advanced Non-small Cell Lung Carcinoma
Brief Title: BAY43-9006 - Phase II Study in Non-Small Cell Lung Carcinoma (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100557
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Results first posted 2010-04-08 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Cancer; Carcinoma, Non-Small Cell Lung
Keywords: NSCLC
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib (Experimental): Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (bid, bis in die) X 28 day cycles
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — BAY43-9006 400 mg bid X 28 day cycles [Continuous treatment for a maximum of 2 years; potential for compassionate use and long term survival follow-up post drug discontinuation.

SUMMARY:
The purpose of the study is to evaluate if BAY43-9006 has an effect on the tumors, how long the effect continues, if the patients receiving BAY43-9006 will live longer.

* If BAY43-9006 has an effect on the quality of life of patients with non-small cell lung cancer.
* If BAY43-9006 helps to slow the worsening of non-small cell lung cancer.
* If BAY43-9006 prevents the growth of, or shrinks non-small cell lung tumors and/or their metastases.

DETAILED DESCRIPTION:
In addition to the key secondary outcome parameters several potential biomarkers were evaluated as exploratory parameters.

Issues on safety are addressed in the Adverse Event section.

The following acronyms and abbreviations were used in the Adverse Event section and Limitations and Caveats section:

* gastrointestinal (GI)
* not otherwise specified (NOS)
* central nervous system (CNS)
* National Cancer Institute Common Terminology Criteria (NCI-CTC)
* Medical Dictionary for Regulatory Activities (MedDRA)
* System Organ Class (SOC)
* interim analysis (IA)

ELIGIBILITY:
Inclusion Criteria:

* Age = 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* Life expectancy of at least 12 weeks at the pre-treatment evaluation
* Patients with metastatic, measurable, histologically or cytologically documented NSCLC (includes squamous, large cell or adenocarcinoma). In case of unique metastatic site, histological confirmation is required in order to ensure proper diagnosis prior to study entry
* Patients must have progressive non-small cell lung cancer (NSCLC)
* No more than 2 prior systemic agent or regimen at least 28 days prior to study entry. (Prior therapy with gefitinib is allowed but not mandatory)
* Patients must be considered appropriate for systemic anti-cancer therapy by the Investigator
* Patients with at least one uni-dimensional measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Adequate bone marrow, liver and renal function, as assessed by the following laboratory:
* Hemoglobin = 9.0 g/dl
* Absolute granulocytes = 1.5 x 10E9/L
* Platelet count = 100 x 10E9/L
* Total bilirubin < 1.5 x the upper limit of normal
* alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer)
* prothrombin time (PT) or International Normalized Ratio (INR) and partial thromboplastin time (PTT) < 1.5 x upper limit of normal (except in patients who are on warfarin or heparin. Patients who receive anti-coagulation treatment with an agent such as warfarin or heparin, prophylactically or therapeutically, will be allowed to participate. For patients on warfarin, close monitoring of at least weekly evaluations will be performed until INR is stable based on a measurement at pre dose, as defined by the local standard of care)
* Serum creatinine = 2.0 x upper limit of normal
* Amylase and lipase < 1.5 x the upper limit of normal

Exclusion Criteria:

* Cardiac arrhythmia requiring anti-arrhythmics (excluding beta-blockers or digoxin), symptomatic coronary artery disease (CAD) or ischemia (myocardial infarction (MI) within the last 6 months) or congestive heart failure (CHF) > New York Heart Association (NYHA) Class II
* Uncontrolled hypertension
* Complete renal shut-down requiring hemo- or peritoneal dialysis
* Mixed histologies
* Active clinically serious infections (> grade 2 on the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0)
* Known history of HIV infection or chronic hepatitis B or C
* Known metastatic brain or meningeal tumors, unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry. A head CT or MRI must be conducted to rule out brain metastasis or meningeal tumors. Also the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable, provided that the dose is stable for one month prior to and following screening radiographic studies)
* History of seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft and bone marrow transplant
* Previous malignancy (except for cervical carcinoma in situ, adequately treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis & T1] or other malignancies curatively treated > 3 years prior to entry)
* Patients with clinically significant bleeding (e.g., gastrointestinal bleeding) within the past month prior to study entry are ineligible
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures (e.g. cervical cap, condom, and diaphragm) during the course of the trial. Oral birth control methods alone will not be considered adequate on this study, because of the potential pharmacokinetic interaction between BAY 43-9006 and oral contraceptives
* Substance abuse, medical, psychological or social conditions that, in the judgment of the investigator, is likely to interfere with the patients participation in the study or evaluation of the study results
* Known allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or could jeopardize the safety of the patient and its compliance in the study, in the investigator's judgment
* Anti cancer chemotherapy, immunotherapy, vaccines or investigational therapy during the study or within 4 weeks of study entry.
* Radiotherapy during the study or within 4 weeks of study entry. Patients must have recovered from radiation-induced toxicity. However, palliative is allowed for local pain control.
* Any surgical procedure within 4 weeks prior to the start of study drug. Autologous and/or allogenic including mini-allogenic bone marrow transplant or stem cell rescue. Use of biologic response modifiers, such as Granulocyte-Colony Stimulating Factor (G-CSF) or Granulocyte macrophage colony-stimulating factor (GM-CSF), during or within 3 weeks of study entry. G-CSF and other hematopoietic growth factors may only be used in the management of acute toxicity, when medically indicated, or at the discretion of the investigator. Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study. Use of St. John's Wort. Use of rifampicin. Prior use of Raf-Kinase inhibitors, MAPK/ERK kinase (MEK) or Farnesyl Transferase Inhibitors. Prior use of Bevacizumab and all other drugs that target vascular endothelial growth factor (VEGF)/ vascular endothelial growth factor receptor (VEGFR). Use of any investigational drug therapy outside of this during or within 4 weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-04; Primary Completion 2005-06 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Houston, Texas, United States
- Großhansdorf, Schleswig-Holstein, Germany

REFERENCES:
- [Result] Blumenschein GR Jr, Reck M, Fossella F, Stewart DJ, Lathia C, Pena C. Plasma biomarkers correlating with clinical outcome in a phase II study of sorafenib in advanced NSCLC. Cancer Biomark. 2011-2012;10(6):287-98. doi: 10.3233/CBM-2012-0253. PMID 22820084
- [Result] Blumenschein GR Jr, Gatzemeier U, Fossella F, Stewart DJ, Cupit L, Cihon F, O'Leary J, Reck M. Phase II, multicenter, uncontrolled trial of single-agent sorafenib in patients with relapsed or refractory, advanced non-small-cell lung cancer. J Clin Oncol. 2009 Sep 10;27(26):4274-80. doi: 10.1200/JCO.2009.22.0541. Epub 2009 Aug 3. PMID 19652055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted in Germany and USA (1 center each) from Apr 2004 to Jun 2005. Recruitment in 2 phases: Interim analysis (IA) to be performed after treatment of 29 patients; final analysis planned after additional 21 patients. Final analysis data cut-off date 30 Jun 2005; safety data collected for the 4 ongoing subjects until 11 Apr 2008.
Pre-assignment Details: 52 of 54 enrolled patients started treatment. The analysis population consisted of 52 subjects for the intent to treat (ITT) and safety analyses and 51 subjects in the evaluable subject analysis (1 had lung metastases from pancreatic cancer).
Period: Overall Study
Arm/Group | Sorafenib
Started | 52
Completed | 52 (Safety data collected for 4 subjects after 30 Jun 2005 until 11 Apr 2008.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib
Number analyzed (Participants) | 52
Age Continuous [Median (Full Range); unit: years] | 62 [26 to 85]
Age, Customized [Number; unit: participants]
  >=65 years | 21
  < 65 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 34
Histology [Number; unit: participants] — Measurable, histologically or cytologically documented stage IV non-small cell lung cancer (NSCLC). Subjects must have had disease progression at the time of study entry and have been treated with at least 1 but no more than 2 prior systemic agents or regimens (including gefitinib).
  participants
    Adenocarcinoma NSCLC | 28
    Large cell carcinoma | 4
    Squamous cell (epidermoid) carcinoma | 16
    Undifferentiated carcinoma | 4

OUTCOME MEASURES:

1. Primary Outcome: Anti-cancer Activity (eg, Percentage of Patients With Confirmed Complete Responses (CR) and Partial Responses (PR) Per RECIST (Response Evaluation Criteria in Solid Tumors) Criteria in Patients With Stage IV Non-small Cell Lung Carcinoma (NSCLC)
Description: CR-disappearance of clinical/radiological tumor evidence (target/nontarget). PR- >=30% decrease in sum longest diameter (LD) of target lesions from BL sum LD. Stable disease (SD)-no shrinkage for PR nor increase for PD. Progressive disease (PD) measurement proven- >=20% increase in sum LD of lesions from smallest sum LD since start or new lesions. Progression by clinical judgement- >clinically meaningful cancer-related deterioration as judged by the investigator.
Time Frame: First patient first treatment until date for last data collection for efficacy for a study period up to 62 weeks. Tumor assessed per RECIST at baseline (BL), every 8 weeks during treatment and at end of treatment.
Population: The analysis population for the intent to treat (ITT) and safety analyses consisted of 52 subjects who received at least 1 treatment and had their disease re-evaluated. 51 subjects were considered evaluable since 1 of the 52 subjects had lung metastases from pancreatic cancer.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 51
percentage of participants
  Complete response + Partial response | 0.0
  Complete response | 0.0
  Partial response | 0.0
  Stable disease | 58.8
  Progressive disease measurement proven | 23.5
  Progression by clinical judgement | 11.8
  Not evaluated | 5.9

2. Secondary Outcome: Duration of Stable Disease
Description: Duration of stable disease was calculated as date of first treatment until date of documented progressive disease (PD) or last observation if subject did not progress. Stable disease (SD) defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Kaplan-Meier methodology, descriptive analysis.
Time Frame: as for outcome 1
Population: The analysis population for the intent to treat (ITT) and safety analyses consisted of 52 subjects who received at least 1 treatment and had their disease re-evaluated. 1 of the 52 subjects had lung metastases from pancreatic cancer and was excluded from analysis. 48 subjects had tumor evaluations post-baseline and were evaluable.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib
Number analyzed (Participants) | 48
days | 103 [58 to 116]

3. Secondary Outcome: Overall Survival
Description: Overall survival was calculated from the date of the first treatment until death of the subject.
  Evaluation by Kaplan-Meier methodology, descriptive analysis.
Time Frame: First patient first treatment until date for last data collection for efficacy for a study period up to 62 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib
Number analyzed (Participants) | 51
days | 205 [151 to 257]

4. Secondary Outcome: Percentage of Subjects With Stable Disease (SD)
Description: Percentage of subjects with stable disease was calculated from date of first treatment until date of documented progressive disease (PD) or last observation if subject did not progress. Stable disease (SD) defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Descriptive summary of subjects with SD.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 51
Percentage of participants | 58.8

5. Secondary Outcome: Change From Baseline of Health-Related Quality of Life (HRQOL) Score Assessed at Cycle 2, Cycle 4, and End of Treatment (EOT)
Description: HRQoL was assessed with the FACT-L questionnaire, a validated instrument for determining lung cancer HRQoL. The 36-item questionnaire includes 4 domains: Physical, functional, emotional, and social/family well-being, and a lung cancer-specific subscale. The FACT-L total score ranges from 1 to 136. Lower scores (negative change from baseline) demonstrate impaired HRQoL.
Time Frame: From first patient first treatment until date of last efficacy data collection (study period up to 62 weeks). HRQoL assessed at baseline (BL), end of treatment Cycles 2 and 4, and at end of treatment
Population: The analysis population for the intent to treat (ITT) and safety analyses consisted of 52 subjects who received at least 1 treatment and had their disease re-evaluated. Of the 52 treated subjects, 50 subjects completed the FACT-L at baseline (screening) and post-treatment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sorafenib
Number analyzed (Participants) | 50
scores on a scale
  Cycle 2 | -4.8 (21.2)
  Cycle 4 | 0.0 (14.4)
  End of treatment | -14.9 (23.2)

ADVERSE EVENTS:
Time Frame: AE data were collected from Apr 2004 to Apr 2008
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 28/52
Other Adverse Events (participants affected / at risk) | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=52)
Hemoglobin (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Cardiac arrythmia - other (Cardiac disorders) | 1
Cardiac general - other (Cardiac disorders) | 6
Hypertension (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Death not associated with ctcae term, disease progression nos (General disorders) | 6
Fatigue (General disorders) | 5
Constitutional symptoms - other (General disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Fistula, GI, esophagus (Gastrointestinal disorders) | 1
GI - other (Gastrointestinal disorders) | 1
Stricture, GI, (Gastrointestinal disorders) | 1
Hemorrhage, GI, upper GI nos (Vascular disorders) | 1
Hemorrhage pulmonary, respiratory tract nos (Vascular disorders) | 1
Hepatobiliary -other (Hepatobiliary disorders) | 2
Pancreatitis (Hepatobiliary disorders) | 1
Infection (documented clinically), lung pneumonia (Infections and infestations) | 2
Dermal change (Blood and lymphatic system disorders) | 1
Edema: limb (Blood and lymphatic system disorders) | 1
Bilirubin (Metabolism and nutrition disorders) | 2
Amylase (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Lipase (Metabolism and nutrition disorders) | 1
Metabolic/lab - other (Metabolism and nutrition disorders) | 1
CNS ischemia (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Mental status (Nervous system disorders) | 1
Neurology - other (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Pain, abdomen nos (Gastrointestinal disorders) | 2
Pain, chest/thorax nos (General disorders) | 1
Pain, head/headache (General disorders) | 1
Pain, other (General disorders) | 1
Pain, neck (General disorders) | 1
Pain, stomach (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Fistula, pulmonary, bronchus (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=52)
Hypertension (Cardiac disorders) | 13
Fatigue (General disorders) | 32
Weight loss (General disorders) | 16
Fever (General disorders) | 12
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 19
Dermatology - other (Skin and subcutaneous tissue disorders) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 12
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11
Diarrhea (Gastrointestinal disorders) | 27
Anorexia (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 11
Infection - other (Infections and infestations) | 12
Dermal change (Blood and lymphatic system disorders) | 14
Pain, other (General disorders) | 19
Pain, chest/thorax nos (General disorders) | 14
Pain, head/headache (General disorders) | 14
Pain, back (General disorders) | 11
Pain, abdomen nos (General disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 27
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 12
Hemoglobin (Blood and lymphatic system disorders) | 3
Hypotension (Cardiac disorders) | 5
Cardiac general - other (Cardiac disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 10
Nail changes (Skin and subcutaneous tissue disorders) | 3
Insomnia (General disorders) | 3
Constitutional symptoms - other (General disorders) | 10
Rigors/chills (General disorders) | 5
Sweating (General disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 4
Heartburn (Gastrointestinal disorders) | 3
Mucositis (clinical exam), oral cavitiy (Gastrointestinal disorders) | 6
GI - other (Gastrointestinal disorders) | 8
Hemorrhage - other (Vascular disorders) | 3
Hemorrhage pulmonary, bronchopulmonary NOS (Vascular disorders) | 3
Hemorrhage pulmonary, nose (Vascular disorders) | 4
Musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 3
Gait/walking (Musculoskeletal and connective tissue disorders) | 3
AST (Metabolism and nutrition disorders) | 4
Creatinine (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Lipase (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Metabolic/lab - other (Metabolism and nutrition disorders) | 6
Mood alteration, anxiety (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 8
Mood alteration, depression (Nervous system disorders) | 6
Neurology - other (Nervous system disorders) | 8
Neuropathy - sensory (Nervous system disorders) | 3
Ocular - other (Eye disorders) | 3
Pain, chest wall (General disorders) | 5
Pain, extremity - limb (General disorders) | 10
Pain, tumor pain (General disorders) | 3
Pain, joint (General disorders) | 6
Pain, muscle (General disorders) | 5
Pain, bone (General disorders) | 3
Pain, neck (General disorders) | 8
Pain, stomach (General disorders) | 9
Pain, throat/pharynx/larynx (General disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes (Respiratory, thoracic and mediastinal disorders) | 6
Urinary frequency (Renal and urinary disorders) | 3
Renal - other (Renal and urinary disorders) | 3

LIMITATIONS AND CAVEATS:
Due to rapid enrollment, no IA (interim analysis) was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less